CLINICAL TRIAL: NCT01805739
Title: Multi Modal Cardiac Imaging Prior Transcatheter Aortic Valve Implantation (TAVI)
Brief Title: Multi Modal Cardiac Imaging Prior Transcatheter Aortic Valve Implantation
Status: Recruiting | Type: Observational
Sponsor: Klinik für Kardiologie, Pneumologie und Angiologie (Other)
Responsible Party: Sponsor-Investigator, Klinik für Kardiologie, Pneumologie und Angiologie, Director Division of Cardiology, Pulmonary Diseases, Vascular Medicine, Heinrich-Heine University, Duesseldorf
Organization: Heinrich-Heine University, Duesseldorf (Other)
Other Study IDs: Multi Modal Cardiac Imaging
Record Dates: First submitted 2013-03-01; First posted 2013-03-06 (Estimated); Last update posted 2020-10-30 (Actual); Status verified 2020-10

CONDITIONS: Aortic Valve Stenosis
Keywords: transcatheter aortic valve implantation; CT; MRI; angiography; echocardiography; rotational C-arm CT
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No

SUMMARY:
Transcatheter aortic valve implantation (TAVI) is an emerging alternative therapy for aortic stenosis for patients ineligible for open heart surgery or at high risk for perioperative complications. Pre-procedural imaging of the aortic root is essential for selection of the correct valve prosthesis and to minimize complications as prosthesis mismatch, possibly subsequent embolization, coronary obstruction, annulus rupture or severe aortic regurgitation.

The aim of the study is to compare the different imaging modalities for aortic root measurements.

Aortic root imaging will be performed prior to TAVI-procedure. The contrast injection will be performed either into the aorta or into the left ventricle. The datasets will be assessed by blinded-independent observers in a multi-planar reconstruction view.

The study will be performed retrospectively (2009-2012) and prospectively starting 2013.

DETAILED DESCRIPTION:
Transcatheter aortic valve implantation (TAVI) is an emerging alternative therapy for aortic stenosis for patients ineligible for open heart surgery or at high risk for perioperative complications. Pre-procedural imaging of the aortic root is essential for selection of the correct valve prosthesis and to minimize complications as prosthesis mismatch, possibly subsequent embolization, coronary obstruction, annulus rupture or severe aortic regurgitation.

The aim of the study is to compare the different imaging modalities for aortic root measurements.

Aortic root imaging will be performed prior to TAVI-procedure. The contrast injection will be performed either into the aorta or into the left ventricle. The datasets will be assessed by blinded-independent observers in a multi-planar reconstruction view.

The study will be performed retrospectively (2009-2012) and prospectively starting 2013.

Substudy: "Real-World Experience with Implantation Depth Optimization according to 2020 Recommendations for Evolut R Self-Expanding Transcatheter Aortic Valve: the Düsseldorf Best Practice Trial." Aortic valve stenosis treated by transcatheter aortic valve replacement (TAVR) is one of the most fast-growing sections in interventional cardiology. The Heart Center Düsseldorf is a high-volume center for treatment of patients suffering of aortic stenosis treated by TAVR, so we have a great interest in further investigation of process optimizing and improvement. Therefore, we will focus on optimization of implantation depth (ID) according to Medtronic®'s best practice recommendations for TAVR deployment in July 2020 regarding new-generation devices Medtronic® CoreValve Evolut. Optimal ID is an important condition for hemodynamic and clinical outcome due to increased risk of paravalvular leakage or even valve embolization in implantation that is located too high, whereas deep implantation is associated with more aortic regurgitation an increased risk of conduction disturbances associated with higher rates of permanent pacemaker implantation. The aim of this single-center observational study is to investigate short-term clinical performance, safety and efficiency outcomes in patients undergoing transfemoral TAVR regarding Medtronic®'s best practice advices of July 2020 for TAVR deployment with CoreValve Evolut.

ELIGIBILITY:
Inclusion Criteria:

* aortic valve stenosis
* screened for TAVI
* written informed consent

Exclusion Criteria:

* unconsciousness, not able to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with aortic valve stenosis screened for TAVI
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2013-01; Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Assessment of diameters of the aortic annulus using the different imaging modalities | baseline
Implantation depth (ID) measured from NCC in fluoroscopic view | baseline

SECONDARY OUTCOMES:
left ventricular contrast injection | baseline
Comparison of pre-procedural TAVI-imaging for the assessment of the left ventricular outflow tract (LVOT). | baseline
mean pressure gradient | baseline
paravalvular aortic regurgitation | baseline
bleeding and vascular access site complications | baseline

OTHER OUTCOMES:
Major Adverse Cardiac Event | 1 month, 3 months and 12 months
Hospitalisation | 1 month, 3 months and 12 months
Mortality | 1 month, 3 months and 12 months
blood samples | 1 month, 3 months and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Malte Kelm, MD, Study Director — Division of Cardiology, Pulmonary Diseases, Vascular Medicine, University Hospital Duesseldorf
Locations (1):
- Division of Cardiology, Pulmonary Diseases, Vascular Medicine, University Hospital Duesseldorf, Düsseldorf, North Rhine-Westphalia, Germany

REFERENCES:
- [Derived] Veulemans V, Heermann J, Adrichem R, Hecht S, Seppelt PC, Hokken TW, Nuis RJ, Abdel-Wahab M, van Mieghem NM, Leistner D, Vorpahl MM, Zeus T. Evidence of bioprosthetic valve dysfunction during three-year follow-up following TAVR. Clin Res Cardiol. 2025 May 12. doi: 10.1007/s00392-025-02630-7. Online ahead of print. PMID 40353875
- [Derived] Quast C, Bonner F, Polzin A, Veulemans V, Chennupati R, Gyamfi Poku I, Pfeiler S, Kramser N, Nankinova M, Staub N, Zweck E, Jokiel J, Keyser F, Hoffe J, Witkowski S, Becker K, Leuders P, Zako S, Erkens R, Jung C, Flogel U, Wang T, Neidlin M, Steinseifer U, Niepmann ST, Zimmer S, Gerdes N, Cortese-Krott MM, Feelisch M, Zeus T, Kelm M. Aortic Valve Stenosis Causes Accumulation of Extracellular Hemoglobin and Systemic Endothelial Dysfunction. Circulation. 2024 Sep 17;150(12):952-965. doi: 10.1161/CIRCULATIONAHA.123.064747. Epub 2024 Jun 5. PMID 38836358
- [Derived] Veulemans V, Maier O, Piayda K, Berning KL, Binnebossel S, Polzin A, Afzal S, Dannenberg L, Horn P, Jung C, Westenfeld R, Kelm M, Zeus T. Factors associated with a high or low implantation of self-expanding devices in TAVR. Clin Res Cardiol. 2021 Dec;110(12):1930-1938. doi: 10.1007/s00392-021-01901-3. Epub 2021 Jun 24. PMID 34165599
- [Derived] Piayda K, Dannenberg L, Zako S, Maier O, Bosbach G, Polzin A, Afzal S, Jung C, Westenfeld R, Kelm M, Zeus T, Veulemans V. Predictors of calcification distribution in severe tricuspid aortic valve stenosis. Int J Cardiovasc Imaging. 2021 Sep;37(9):2791-2799. doi: 10.1007/s10554-021-02248-6. Epub 2021 Apr 20. PMID 33877483
- [Derived] Veulemans V, Maier O, Bosbach G, Hellhammer K, Afzal S, Piayda K, Polzin A, Jung C, Westenfeld R, Mehdiani A, Lichtenberg A, Kelm M, Zeus T. Impact of Combined "CHADS-BLED" Score to Predict Short-Term Outcomes in Transfemoral and Transapical Aortic Valve Replacement. J Interv Cardiol. 2020 Dec 18;2020:9414397. doi: 10.1155/2020/9414397. eCollection 2020. PMID 33380924
- [Derived] Piayda K, Hellhammer K, Veulemans V, Sievert H, Gafoor S, Afzal S, Hennig I, Makosch M, Polzin A, Jung C, Westenfeld R, Kelm M, Zeus T. Navigating the "Optimal Implantation Depth" With a Self-Expandable TAVR Device in Daily Clinical Practice. JACC Cardiovasc Interv. 2020 Mar 23;13(6):679-688. doi: 10.1016/j.jcin.2019.07.048. Epub 2019 Dec 11. PMID 31838114
- [Derived] Veulemans V, Zeus T, Kleinebrecht L, Balzer J, Hellhammer K, Polzin A, Horn P, Blehm A, Minol JP, Kropil P, Westenfeld R, Rassaf T, Lichtenberg A, Kelm M. Comparison of Manual and Automated Preprocedural Segmentation Tools to Predict the Annulus Plane Angulation and C-Arm Positioning for Transcatheter Aortic Valve Replacement. PLoS One. 2016 Apr 13;11(4):e0151918. doi: 10.1371/journal.pone.0151918. eCollection 2016. PMID 27073910
- [Derived] Balzer JC, Boering YC, Mollus S, Schmidt M, Hellhammer K, Kroepil P, Westenfeld R, Zeus T, Antoch G, Linke A, Steinseifer U, Merx MW, Kelm M. Left ventricular contrast injection with rotational C-arm CT improves accuracy of aortic annulus measurement during cardiac catheterisation. EuroIntervention. 2014 Jul;10(3):347-54. doi: 10.4244/EIJV10I3A60. PMID 24755302